CLINICAL TRIAL: NCT06145347
Title: Correlation Between the Preoperative N-terminal Pro-B-type Natriuretic Peptide and Acute Kidney Injury After Abdominal Surgery: a Single Center Retrospective Cohort Study Based on ERAS Database
Brief Title: Correlation Between Preoperative NT-proBNP and Postoperative AKI
Status: Completed | Type: Observational
Sponsor: Xijing Hospital (Other)
Responsible Party: Principal Investigator, Chong Lei, MD & phD, Principal investigator, Head of Anesthesia Clinical Research Center, Xijing Hospital, Xijing Hospital
Other Study IDs: KY-20232265-F-1
Record Dates: First submitted 2023-09-14; First posted 2023-11-24 (Actual); Last update posted 2024-08-16 (Actual); Status verified 2024-08

CONDITIONS: Acute Kidney Injury
Keywords: NT-proBNP; AKI; ERAS; abdominal surgery
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Acute kidney injury group: Patients developed acute kidney injury.
- Non-Acute kidney injury group: Patients didn't develope acute kidney injury.

SUMMARY:
Accurate preoperative AKI risk prediction is of great significance for improving patient outcomes. The use of preoperative NT-proBNP can provide a more precise assessment of the body's fluid load status, guide intraoperative and postoperative fluid management, and thus reduce fluid related postoperative complications. Given the potential association between ERAS and increased postoperative AKI, we hypothesize that preoperative NT-proBNP may be associated with the development of postoperative AKI in ERAS, and can improve the prediction of AKI beyond traditional clinical risk factors. This study aims to validate this hypothesis and provide evidence for using NT-proBNP to assess AKI risk before non cardiac surgery. Improve the predictive ability of clinical predictive models and optimize ERAS protocols to prevent postoperative AKI.

DETAILED DESCRIPTION:
Acute kidney injury (AKI) refers to a rapid decrease in glomerular filtration rate. Postoperative AKI refers to AKI that occurs within 7 days after surgery and is one of the serious perioperative complications in surgical patients. The incidence of postoperative AKI reported in different studies ranges from 2% to 39%, with the incidence of AKI after major abdominal surgery reaching as high as 13.4%. Postoperative AKI is associated with poor prognosis of patients, including increased incidence rate of chronic kidney disease, short-term and long-term mortality, prolonged hospitalization and increased medical costs. The data of patients admitted to the intensive care unit after surgery shows that the 10-year survival rate of patients with postoperative AKI is significantly reduced. Early identification of high-risk patients with postoperative AKI is a prerequisite for developing strategies to improve or prevent perioperative kidney injury. In the past decade, preoperative risk prediction models for AKI after non cardiac surgery, such as the SPARK index, have been developed. However, due to the fact that these models mainly rely on medical and medication history, and rarely use objective biomarkers other than glomerular filtration rate, the predictive ability of AKI prediction models currently used in clinical practice is limited.

The occurrence of AKI is related to oxidative stress, cell apoptosis, inflammatory stimulation, and renal ischemia-reperfusion injury caused by insufficient capacity or overload. A randomized clinical trial of 350 people demonstrated that target directed fluid infusion can reduce the occurrence of acute kidney injury. The level of N-terminal B-type natriuretic peptide (NT proBNP) has been proven to accurately reflect the current intravascular fluid balance, without being affected by the hormone axis. Arkom et al. found that NT proBNP can predict the volume load of dialysis patients. In the early stage of pancreatectomy recovery, serum NT proBNP can provide better assessment of intravascular volume compared to BUN/CRN ratio, and BNP levels in patients in the monitoring room are parallel to changes in humoral resuscitation. These data indicate that NT proBNP levels can be used to guide postoperative fluid resuscitation and management.

When myocardial cells are subjected to pressure/stretching stimulation, NT proBNP is produced by the precursor of B-type natriuretic peptide, which is considered to represent the severity of left ventricular dysfunction and can better reflect potential hemodynamic changes and evaluate perioperative risk in surgical patients. NT proBNP is mostly cleared by the kidneys, and recent studies have linked it to the risk of postoperative AKI. Previous studies have reported that the optimal critical value of NT-proBNP in patients with heart failure is influenced by renal dysfunction, and NT-proBNP is significantly elevated in end-stage renal failure patients. It suggests that it may reflect the state of renal function to some extent. The preoperative concentration of NT-proBNP in patients with AKI after non cardiac surgery is significantly higher than that in patients without AKI. In cardiac surgery, an increase in NT-proBNP before surgery is an independent risk factor for postoperative AKI. However, to date, there has been no risk assessment application of NT-proBNP in the non cardiac surgical population.

Postoperative Accelerated Rehabilitation (ERAS) refers to the application of a series of evidence-based and multidisciplinary perioperative optimization measures aimed at reducing the occurrence of complications, promoting rapid recovery of patients, controlling inflammation, reducing stress reactions, and applying evidence-based medicine. Although ERAS brings improvement in patient prognosis, the positive fluid balance caused by ERAS and the use of NSAIDs may lead to damage to renal function. A retrospective study by Patrick S team demonstrated that ERAS is an important risk factor for postoperative AKI. Steven McClane team also found a significant increase in postoperative AKI in colorectal surgery patients who implemented ERAS strategy through propensity score matching.

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 years
2. undergoing elective surgery
3. Have a history of NT-proBNP and creatinine testing within 7 days before surgery

Exclusion Criteria:

1. Patients undergoing chronic peritoneal or hemodialysis treatment; patients who have undergone kidney transplantation; preoperative serum creatinine levels>4.5mg/dL (400 μ Mol/L) or end-stage renal disease patient (defined as glomerular filtration rate<15ml • min-1 • 1.73m-2)
2. Organ transplantation surgery
3. Pregnant patients
4. Surgical duration<1 hour

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with normal renal function undergoing elective abdominal surgery
Sampling Method: Non-Probability Sample
Enrollment: 629 (Actual)
Dates: Start 2023-07-10 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
Incidence of AKI assessed by KDIGO 2012 (Kidney Disease: Improving Global Outcomes) | 1 week
  Postoperative incidence of AKI, serum creatinine increases≥ 0.3mg/dL (≥ 26.5 μ Mol/L) within 48 hours, or the serum creatinine increases to 1.5 times or more of the baseline value within 7 days.

SECONDARY OUTCOMES:
AKI grading assessed by KDIGO 2012 (Kidney Disease: Improving Global Outcomes) | 1 week
  Postoperative AKI grading, KDIGO stage 1 AKI is defined as an increase in serum creatinine of 1.5-1.9 times the baseline value or an increase of ≥ 0.3mg/dL (26.5 μ Mol/L); KDIGO stage 2 AKI: serum creatinine increased to 2-2.9 times the baseline value; KDIGO stage 3 AKI is defined as an increase in blood creatinine to a 3-fold baseline value or 4mg/dL (353.6 μ Mol/L or above, or initiate renal replacement therapy.
Morbidity | 4 week
  Total postoperative complication

CONTACTS AND LOCATIONS:
Overall Officials: Hailong Dong, Study Chair — Xijing Hospital
Locations (1):
- Xijing Hospital, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ojo B, Campbell CH. Perioperative acute kidney injury: impact and recent update. Curr Opin Anaesthesiol. 2022 Apr 1;35(2):215-223. doi: 10.1097/ACO.0000000000001104. PMID 35102042
- [Derived] Zhang Z, Zheng Z, Nie H, Dong H, Lei C. Association between the preoperative N-terminal pro-B-type natriuretic peptide and acute kidney injury in gastrointestinal surgery patients managed with enhanced recovery strategy: a retrospective cohort study. Perioper Med (Lond). 2025 Apr 22;14(1):45. doi: 10.1186/s13741-025-00528-6. PMID 40264198